CLINICAL TRIAL: NCT00573638
Title: The Effects of the Xal-Ease Delivery Aid Device on Patient Compliance With Xalatan Eye Drops
Brief Title: Effects of Xal-Ease on Patient Compliance With Xalatan
Acronym: Xal-Ease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Michelle Christiano, Medical College of Georgia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-02-266; Guarantor or CPI # 002533552
Record Dates: First submitted 2007-12-07; First posted 2007-12-14 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma
Keywords: glaucoma; compliance; eye drops; deliver aid; Patients could range anywhere from 40 to 80 years old; Patients must have diagnosis requiring treatment with Xalatan.; Patients will be male or female and from any racial/ethnic background.
MeSH Terms: conditions — Glaucoma; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Xal-Ease device to be used with Xalatan eye drops — This intervention is a drop instillation guide to be used in conjunction with the FDA approved Xalatan eye drop.

SUMMARY:
The study hypothesis is that the Xal-Ease with increase patient compliance with XALATAN

ELIGIBILITY:
Inclusion Criteria:

* 40 to 80 years old
* Diagnosis warranting treatment with Xalatan eye drops.
* ambulatory and well functioning

Exclusion Criteria:

* non-ambulatory
* less than 40 or greater than 80 years old
* Not using Xalatan eye drops

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-02; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is compliance with the medication XALATAN using and not using the Xal-Ease delivery aid for their glaucoma treatment. | six months

SECONDARY OUTCOMES:
To determine if any of the other factors mentioned in the survey affect compliance to their medical regimen | six months
To see whether or not the Xal-Ease device helps patients conserve medication. ie - aids in drops not distilled in the eye. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian D. Nilson, MD, Principal Investigator — Augusta University
Locations (1):
- Medical College of Georgia Health Inc, Augusta, Georgia, United States